CLINICAL TRIAL: NCT01105351
Title: Effect of Mild Increase in Folic Acid Intake on the Distribution of Folate Forms in Relation to a Common Polymorphism in One Folate Catabolising Enzyme
Brief Title: Effect of Folic Acid on Primary Folate Forms in Relation to MTHFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Rima Obeid, Prof. Dr., Universität des Saarlandes
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Folate Forms MTHFR
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: the Effect of MTHFR C677T on Folate Metabolism
Keywords: Folate; MTHFR; Homocysteine
MeSH Terms: interventions — Folic Acid; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- folic acid plus B6 and B12 (Active Comparator): folic 400 µg plus vitamin B12 plus B6
  Interventions: Dietary Supplement: folic acid plus B6 and B12
- Folic acid (Placebo Comparator): folic acid alone
  Interventions: Dietary Supplement: folic acid

INTERVENTIONS:
Dietary Supplement: folic acid plus B6 and B12 — folic acid 400 µg plus vitamin B12 plus B6
  Other Names: no further names
  Arms: folic acid plus B6 and B12
Dietary Supplement: folic acid — folic acid 400 µg
  Other Names: folic acid alone
  Arms: Folic acid

SUMMARY:
The common polymorphism in MTHFR gene (C677T) has a significant effect on (6S)-5-CH3-H4folate after folic acid supplementation. For example, post supplementation differences in (6S)-5-CH3-H4folate between CC and TT are above 30%.

DETAILED DESCRIPTION:
The investigators aim to test the effect of low doses of folic acid with or without B6 and B12 on folate forms in relation to polymorphisms in folate catabolising enzymes in elderly people. Our hypothesis is that differences in folate forms after folic acid supplementation might be due to polymorphisms in folate catabolising enzymes. Therefore, folic acid might be retained by people with certain genotypes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age > 65 years.

Exclusion Criteria:

* Renal dysfunction
* Recent stroke, or coronary event (within the last 3 months)
* Current cancer treatment
* Antifolate (e.g. methotrexate) treatment
* Ileum resection
* Current B-vitamin supplement
* Epilepsy medications
* Megaloblastic anemia or other indications for treatment with high doses of folate or vitamin B12.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
blood metabolic markers | 18 months
  we will measure primary folate forms after folic acid supplement

CONTACTS AND LOCATIONS:
Overall Officials: Rima Obeid, PhD, Principal Investigator — Department of Clinical Chemistry, University of Saarland
Locations (1):
- University of Saarland, Homburg, Saarland, Germany

REFERENCES:
- [Result] Obeid R, Kirsch SH, Dilmann S, Klein C, Eckert R, Geisel J, Herrmann W. Folic acid causes higher prevalence of detectable unmetabolized folic acid in serum than B-complex: a randomized trial. Eur J Nutr. 2016 Apr;55(3):1021-8. doi: 10.1007/s00394-015-0916-z. Epub 2015 May 6. PMID 25943647